CLINICAL TRIAL: NCT00830492
Title: Comparisin CC/Gonadotropin/GnRH Antagonist and Gonadotropin/GnRH Agonist in IVF Outcome.
Brief Title: Clomiphene Citrate (CC)/Gonadotropin/Gonadotropin Releasing Hormone (GnRH) Antagonist Versus Gonadotropin/GnRH Agonist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yazd Research & Clinical Center for Infertility (Other)
Responsible Party: Mohammad Ali karimzadeh, yazd research and clinical center for IVF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YazdRCCI1388
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Ovarian Stimulation
Keywords: clomiphene citrate; GnRH agonist; GnRH antagonist; in vitro fertilization; clinical pregnancy; pregnancy
MeSH Terms: interventions — Clomiphene; High-Energy Shock Waves; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Buserelin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): In group A (n=100), the patients were stimulated conventional. They desensitized with buserelin (suprefact, Aventis, Frankfurt, Germany) 500µg subcutaneously (S.C.) everyday for menstrual cycle 21, until the baseline evaluation, which takes place in the first few days of menstruation. If baseline levels of estradiol (<50 pg/ml ) had been achieved, then the dose of buserelin would be reduced to 250µg and ovarian stimulation would commence with 150-225 IU recombinant FSH (r_FSH) (Gonal F, Serono, Aubnne, Switzerland) S.C.
  Interventions: Procedure: Ultrasound; Drug: buserelin; Drug: rFSH
- clomiphen/gonadotropin/GnRH antagonist (Experimental): Patients in group B ( n=100 ) were stimulated clomiphene citrate ( ) 100 mg from cycle day three through seven and continuous gonadotropin stimulation with of r_FSH 75 IU daily from cycle day 5. Ultrasound in two group was performed on 8 cycle day. In group B 0.25 mg GnRH antagonist (Ganirelix , Organon ,Netherland ) daily was started with dominant follicle ≥14mm and in this day 75 IU human menopoasl gonadotropin (HMG) (Menogon, ferring, pharmacenticals , Germany ) increased to the initial gonadotropin . LH assessment on the day of starting antagonist was performed and if LH was >15 IU/L , cycle was cancelled. Human chorionic gonadotropin 10000 IU ((pregnyl, Organon, Oss, the Netherlands ) was given when 1 to 3 follicles reached 18 mm
  Interventions: Drug: clomiphene citrate; Procedure: Ultrasound; Drug: GnRH antagonist; Drug: gonadotopin (HMG)

INTERVENTIONS:
Drug: clomiphene citrate — 100 mg from cycle day 3 through 7
  Arms: clomiphen/gonadotropin/GnRH antagonist
Procedure: Ultrasound — cycle day 8
Drug: GnRH antagonist — Daily, started with dominant follicle greater than 14 mm (Ganirelix , Organon, Netherlands).
  Arms: clomiphen/gonadotropin/GnRH antagonist
Drug: gonadotopin (HMG) — 75 IU human menopausal gonadotropin (Menogon, ferring, pharmacenticals , Germany)
  Arms: clomiphen/gonadotropin/GnRH antagonist
Drug: buserelin — Buserelin (suprefact, Aventis, Frankfurt, Germany) 500µg subcutaneously (S.C.) everyday for menstrual cycle 21, until the baseline evaluation, which takes place in the first few days of menstruation. If baseline levels of estradiol (<50 pg/ml ) had been achieved, then the dose of buserelin would be reduced to 250µg.
  Arms: 2
Drug: rFSH — 150-225 IU recombinant FSH (r_FSH) (Gonal F, Serono, Aubnne, Switzerland) S.C.
  Arms: 2

SUMMARY:
Objective: To compare the efficacy of using mild ovarian stimulation protocol and conventional stimulation protocol in IVF outcome.

Design: Prospective randomized trial

Setting: University IVF setting. Patient(s): The study compromised a total 200 subinfertile couple that women had regulary menstruation.

Intervention(s): Patients were randomized to treatment clomiphene citrate, gonadotropin and GnRH antagonist (100 patients) or GnRH agonist and gonadotropin ( 100 patients).

Main outcome measure: Clinical pregnancy rate.

Key Words: clomiphene citrate, GnRH agonist, GnRH antagonist, in vitro fertilization, pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* female patient age 18-35 years, presence of a regular and proven ovulatory menstruation cycle with a length of 26-35 days
* basal FSH <10 IU/L and body mass index (BMI) of 18-30 (kg/m²)
* Indication for IVF were unexplained infertility, mild male factor, tubal factor, early stage endometriosis and cervical factor

Exclusion Criteria:

* patient requiring ICSI

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 2 weeks
ovarian stimulation safety | 3weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yazd Research and Clinical Center For Infertility, Yazd, Yazd Province, Iran